CLINICAL TRIAL: NCT04977856
Title: Efficacy and Cost-effectiveness of Internet-delivered Cognitive Behavior Therapy for Adolescents with Mild to Moderate Depression: a Randomized Controlled Trial of Guided and Self-guided ICBT Vs. Treatment As Usual
Brief Title: Efficacy and Cost-effectiveness of Internet-delivered CBT for Adolescents with Depression
Acronym: IDA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0859
Record Dates: First submitted 2021-07-13; First posted 2021-07-27 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Single-blind parallel-group randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: Assessors conducting post- and follow-up assessments will be blind to treatment allocation, for the full duration of the trial. The outcome measures are identical for both groups, ensuring that the assessors remain blind. At each follow-up assessment, participants will be reminded by their assessor to not reveal their arm allocation. To measure blinding integrity, all assessors will record whether the participating families inadvertently reveal their group allocation, and subsequently guess each participant's treatment allocation at each assessment point and motivate their choice. The blinding will be broken after the trial's final participant has finished his/her 3-month follow-up assessment (primary endpoint). The trial will end when the trial's final participant has finished his/her 3-month follow-up assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Guided ICBT (Experimental): Participants in guided ICBT will receive internet-delivered CBT with therapist support. The treatment consists of 8 online modules with interactive features such as videos and illustrations, delivered over a maximum of 10 weeks. The main treatment focus is behavioral activation. The adolescent and the caregiver are provided with their own separate programs and login to the treatment platform. The caregiver's program also consists of 8 chapters, including psychoeducation about depression and how to support their adolescent in treatment. The adolescents and caregivers have regular contact with a personal assigned therapist via written text messages in the platform. Participants are typically in contact with their therapist several times a week. The adolescent and caregiver can continue to access all treatment modules for the whole follow-up period (3 months), but without therapist-support.
  Interventions: Behavioral: Behavioral activation (BA)
- Self-guided ICBT (Experimental): The self-guided arm is identical to the guided arm, however without the therapist support. To ensure patient safety, there will be clear instructions to the patients and primary caregivers on how to get in contact with the study team in case of acute problems, and there will be clinical routines to detect and manage deterioration or suicidal tendencies.
  Interventions: Behavioral: Behavioral activation (BA)
- Treatment as usual (TAU) (Active Comparator): Participants randomized to TAU, will be referred to the local CAMH's or primary care unit for children and youths and will be free to receive any treatment, either psychosocial, medical, or a combination of both. The content of TAU and the treatment techniques used will be monitored.
  Interventions: Other: Regular care within primary or secondary mental health care for children

INTERVENTIONS:
Behavioral: Behavioral activation (BA) — The main goal of the BA is to increase engagement in values-based activities and decrease avoidant behaviors that serve to maintain depression. The adolescent will learn about depression, how behavioral activations works, monitor their own activities, plan and do more values-based activities and deal with obstacles to getting in touch with positive reinforcement, such as avoidance behaviors.
  Arms: Guided ICBT; Self-guided ICBT
Other: Regular care within primary or secondary mental health care for children — Regular care (supportive therapy, waitlist, psychological treatments, drugs, or a combination of different interventions)
  Arms: Treatment as usual (TAU)

SUMMARY:
Adolescent depression is a prevalent and impairing condition that can be effectively treated with Cognitive Behavior Therapy (CBT). However, a majority of adolescents do not have access to CBT. Internet-delivered CBT (ICBT) has been suggested as a way to increase availability to effective psychological treatments. Yet, the research on ICBT for adolescents has been lagging behind significantly.

The overall aim of this research project is to increase the availability of evidence-based psychological treatments for adolescents with depression by developing and evaluating internet-delivered Cognitive Behavior Therapy (ICBT) for this target group. The main objectives are to establish the efficacy, cost-effectiveness, and long-term effects of the guided and self-guided ICBT for adolescents with mild to moderate depression in a randomized controlled trial (RCT) with three-arms; guided ICBT (with therapist-support) and self-guided ICBT (without therapist-support) vs treatment as usual (TAU).

DETAILED DESCRIPTION:
Primary and secondary objectives

Primary objective:

1. To determine the clinical efficacy of Guided and Self-guided ICBT for depression for reducing depressive symptom severity (as measured by the CDRS-R (27) in adolescents with mild and moderate major depressive disorder (MDD), compared with an active control intervention (treatment as usual within primary or secondary child and adolescent mental health care). The primary endpoint is the follow-up 3 months post-treatment.

Secondary objectives:

1. To establish the 12-month durability of the treatment effects.
2. To conduct a health-economic evaluation of guided ICBT for depression and self-guided ICBT for depression, compared with TAU, from multiple perspectives, both in the short term (primary endpoint) and the long term (12-month follow-up).
3. To investigate potential mediators behind a potential treatment effect of ICBT.

Research questions:

1. Is guided and self-guided ICBT more efficacious than TAU in regard to the reduction of depressive symptoms?
2. Is guided and self-guided ICBT more cost-effective than TAU?
3. Is self-guided ICBT more cost-effective than guided ICBT?
4. Are the therapeutic gains of ICBT maintained long term (i.e., 1 year after the intervention)?
5. Do changes in activation and avoidance (BADS) mediate changes at post-treatment in self-reported depressive symptoms (QIDS-A-17) in adolescents receiving ICBT (with or without therapist support), but not in the control group (treatment as usual)?

ELIGIBILITY:
Inclusion Criteria:

* 13-17 years of age,
* A diagnosis of mild to moderate MDD based on the DSM-5,
* Willing to be randomized to either of the three treatment arms,
* Basic proficiency in Swedish, both adolescent, and a participating caregiver
* Regular access to a desktop, laptop computer connected to the internet, as well as a mobile phone,
* If using medication with antidepressants, central stimulants, or neuroleptics it has to be unchanged at least 6 weeks prior to inclusion, and
* A minimum of one caregiver that is able to co-participate in the treatment.

Exclusion Criteria:

* The presence of psychiatric problems requiring immediate treatment (e.g., high risk of suicide, psychosis, severe self-injury, bipolar disorder, clinical eating disorder, alcohol/substance abuse),
* Social problems requiring immediate action (e.g., ongoing abuse in the family, high and prolonged absence from school);
* Previous psychological treatment for MDD (CBT, interpersonal psychotherapy (IPT), or BA) for a minimum of at least 3 sessions within the last 12 months prior to assessment.
* Current use of benzodiazepines.
* Ongoing psychological treatment for any psychiatric disorder.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 215 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in clinician-rated depressive scores on Children's Depression Rating Scale - Revised (CDRS-R) | week 0, week 10, at 3 and 12 months follow-up
  CDRS-R is a semi-structured clinician interview, assessing level of depressive symptomatology. Total range is 17-113, with higher values representing a worse outcome.

SECONDARY OUTCOMES:
Clinical Global Impression Scale - Severity (CGI-S) | week 0, week 10, at 3 and 12 months follow-up
  CGI-S was developed to assess how mentally ill a specific patient compared to a particular patient population (e.g. with major depressive disorder) at a certain time. It consists of a single item rated on a seven-point scale ranging from 1="no symptoms" to 7="extreme symptoms".
Clinical Global Impression - Improvement (CGI-I) | week 10, at 3- and 12 months follow-up
  CGI-I is developed to assess improvement of psychiatric symptoms for a specific patient compared to baseline. It consists of a single item rated on a seven-point scale ranging from 1="very much improved" to 7="very much worse".
Children's global assessment scale (CGAS) | week 0, week 10, at 3 and 12 months follow-up
  The CGAS is a single item 1-100 scale that integrates psychological, social, and academic functioning in children as a measure of psychiatric disturbance. Higher values represent a better outcome.
Internet Intervention Patient Adherence Scale (iiPAS) | Week 10
  The iiPAS is a clinician-rated measure of patient adherence to internet-delivered behavioral interventions (38) with 5 items rated on a 0 to 4 Likert scale with total score ranging from 0 to 20, where 0 indicates no adherence and 20 perfect adherence. The scale covers client's work pace, engagement, communication with the therapist, motivation for change, and login frequency. The iiPAS has demonstrated excellent internal consistency and good construct validity as well as a strong association with objective measures of patient activity in ICBT(38). For participants in the self-guided group, we will use an adapted version excluding item 3 since communication with therapist is not applicable, and a research assistant will make the rating at post-treatment.
Anhedonia Scale for Adolescents (ASA) | week 0, week 10, at 3 and 12 months follow-up
  The ASA is an adolescent specific measure of anhedonia with 14 items with a four graded-scale from 0 (never) to 3 (always), ranging from 0 to 42 points. A higher score indicates more anhedonia. The ASA has high test-retest reliability and good convergent validity with standardized measures of depression.
Affective Reactivity Index (ARI) | week 0, week 10, at 3 and 12 months follow-up
  The ARI is a measure of irritability, consisting of six items with a three graded scale and one item on impairment due to irritability, ranging from 0 to 12 points with higher scores indicating a worse outcome. The ARI has demonstrated an excellent internal consistency and differentiates cases from controls in a clinic a community sample.
Behavioral activation of Depression Scale - short form (BADS-S) | week 0, weekly during treatment (week 1 to week 10), at 3- and 12 months follow-up
  The BADS-S is designed to track changes in proposed mediators of behavioral activation, e.g. activation and avoidance. Total range is from 0-54 with higher values indicating higher degree of activation and lower degree of avoidance. Changes during treatment in proposed mediators of behavioral activation on the BADS-S will be reported for the ICBT interventions.
Concomitant interventions | Week 10 and 3- and 12-months follow-up assessments.
  To assess if the adolescent has received other psychological treatments during the trial period, the adolescents answer questions about other potential psychological treatments they have received apart from the interventions included in the trial.
The Client Satisfaction Questionnaire-8 (CSQ-8) - adolescent and parent version | week 10
  The CSQ-8 is an 8-item self-rated 4-point scale, measuring different aspects of satisfaction with treatment, e.g. perception of quality of treatment, if the treatment adequately addressed their needs and overall satisfaction. Total range is 8 to 32, with higher values indicating higher satisfaction. Mean in total satisfaction scores on the CSQ-8 for each treatment group at end of treatment and at follow-up will be reported.
Insomnia Severity Index (ISI) | week 0, week 10, and at 3- and 12 months follow-up
  ISI, a brief screening measure of insomnia, a seven-item scale ranging from 0 to 28 points, with higher values representing a worse outcome.
Kidscreen-10 Index - adolescent and parent version | week 0, week 10, at 3- and 12-months follow-up
  Kidscreen-10 assess the adolescents' general health-related quality of life. Total range from 10-50, with higher values indicating better health-related quality of life.
Need for further treatment - adolescent and parent version | at 3 months follow-up
  Investigate whether the participant considers her/himself in need of further treatment for her/his depression. The scale ranges from 0 (no need for more treatment) to 4 (great need for more treatment) where higher scores indicate a worse outcome.
Negative Effects Questionnaire (NEQ-20) - adolescent and parent version | Week 10 and 3 months follow-up
  NEQ-20 investigates participants' negative effects of psychological treatments. Total range is 0-80, with higher values representing a worse outcome.
The Revised Children's Anxiety and Depression Scale, short (RCADS-S) -adolescent and parent version | week 0, week 10, 3- and 12 months follow-up
  The RCADS-S, a shortened version of the Spence Child Anxiety Scale, is a child and parent self-report measure of anxiety- and depression-related psychopathology. Only the anxiety subscales are administered in this study since depressive symptoms are measured thoroughly by other measures. Total range is 0-45, with higher values representing a worse outcome.
Quick Inventory of Depressive Symptomatology, 17 items (QIDS-17) - adolescent and parent version | week 0, weekly from week 1 to week 10, at 3- and 12 months follow-up
  The QIDS-17 covers the nine symptoms defined in the Diagnostic Statistical Manual of Mental Disorders (DSM-5) of depression rated in a scale from 0 (none) to 3 (highest) with a sum-range of 0-27. A total score of 6-10 indicates mild depression, 11-15 moderate, 16-20 severe and 21 and above very severe. Response is defined as a reduction by half of the initial score on QIDS-17. Remission is defined as below 6 points on QIDS-17. The QIDS-17 is a very reliable measure and most discriminating at moderate levels of depression.
Work and Social Adjustment Scale, youth version (WSAS-Y) - adolescent and parent version | week 0, week 10, 3- and 12 months follow-up
  WSAS-Y is a parent- and adolescent-rated scale of impaired functioning in school, everyday life, friends and social life, recreation and hobbies and family and close relationships. The scale generates a global score ranging from 0 to 40, with higher scores indicating greater impairment.
The Expressed Emotion Adjective Checklist (EEAC) | week 0, week 10, 3- and 12 months follow-up
  The EEAC is a validated self-rated questionnaire of the caregiver's positive and negative emotions directed towards the adolescent. The EEAC include 20 adjectives (each scored 1-8 where 1 indicates never and 8 always).
Trimbos Questionnaire for Costs associated with Psychiatric Illness (TiC-P) | week 0, week 10, at 3- and 12 months follow-up
  The TiC-P assess healthcare and societal resource use, including for example items on healthcare resource use, medications, school absenteeism, and parental productivity loss. In the present study no health economic evaluations will be conducted. Rather this instrument is included to gain feasibility data in preparation of a planned larger randomized controlled study. Therefore, no data on TiC-P will be reported in this trial.
  The TiC-P assess healthcare and societal resource use, including for example items on healthcare resource use, medications, school absenteeism, and parental productivity loss.
Treatment credibility - adolescent and parent version | week 3
  Four qualitative questions about treatment credibility will be administered at week 3, asking how well the treatment suits adolescents with depression, how much they believe this treatment will help him/her, if and to what extent they would recommend this treatment to a friend with depression and how much improvement they expect from the treatment. Each item is scored on a 5-point Likert scale, from 1 to 5. The scale ranges from 4 to 20 points, where a higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Serlachius, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- BUP Internetbehandling, BUP Forsknings- och utvecklingscentrum i Stockholm, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersson R, Vigerland S, Lenhard F, Ahlen J, Bottai M, Mataix-Cols D, Serlachius E. Single-blinded, randomised, parallel-group, controlled trial comparing the efficacy and cost-effectiveness of therapist- and self-guided internet-delivered behavioural activation versus treatment as usual for adolescents with mild to moderate depression: study protocol. BMJ Open. 2024 Oct 15;14(10):e083507. doi: 10.1136/bmjopen-2023-083507. PMID 39414268